CLINICAL TRIAL: NCT04242693
Title: Effectiveness of Self-Monitoring and Goal Setting on Improving Consumption of Red/Orange Vegetables Among Undergraduate Students: A Pre-Posttest Experiment
Brief Title: Mobile Goal-setting Intervention to Improve Vegetable Intake Among Young College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Trishnee Bhurosy, PhD, Postdoctoral Fellow, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1711199200
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either an experimental or a control group after they completed a preliminary questionnaire.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group were asked to count the number of times they ate any red/orange vegetables and set a goal to eat one more time the next day over three days.
  Interventions: Behavioral: Mobile goal-setting intervention
- Control Group (No Intervention): The control group uploaded photos and/or descriptions of their meals only. They did not self-monitor their vegetable intake nor set a goal to eat more.

INTERVENTIONS:
Behavioral: Mobile goal-setting intervention — This intervention applied two constructs from the goal setting theory-self-monitoring and goal setting. Briefly, all participants were asked to take photos of all their meals and upload them with descriptions to an online platform. The participants in the experimental group were taken through two additional processes that represented these two constructs. Self-monitoring was operationalized by asking those in the experimental group to count the number of times they ate red/orange vegetables using a counting checklist. Goal setting was operationalized as asking them to set a goal to eat red/orange vegetables one more time tomorrow.
  Arms: Experimental Group

SUMMARY:
This study used a two-group pre-posttest experimental design. After completing a background survey, participants used their smartphones to uploaded photos and/or descriptions of their meals to an online platform for three days. In addition, those in the intervention group were asked to use a checklist to count the number of times they ate red/orange vegetables and to set a goal to eat one more time the next day. The dependent variable was a measure of eating behavior-an estimate (number of times/day) of red/orange vegetable intake on that day based on review of uploaded photos and descriptions. Those in the intervention group, who were asked to use a checklist to count their red/orange vegetable intake and set a goal to eat one more the next day, improved their vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Undergraduate at the university
* Currently lived in a dorm
* Owned a smartphone
* Had internet access on their smartphone

Exclusion Criteria:

* Already part of a study to change their eating behaviors

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Red/orange vegetable intake | Three days
  Number of times participants consumed red/orange vegetables

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Middlestadt, PhD, Study Chair — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data can be shared upon reasonable request. There are identifiers with respect to photos and descriptions provided by participants in the study and these are confidential.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is stored in a secured storage device with the Principal Investigator. The data without any identifiers can only be shared upon a reasonable request.
Access Criteria: Interested individuals should contact the Principal Investigator via email.